CLINICAL TRIAL: NCT04648800
Title: A Multi-centre, Randomised, Double-blind, Placebo-controlled Phase III Clinical Trial Evaluating the Effect of BCG Vaccination on the Incidence and Severity of SARS-CoV-2 Infections Among Healthcare Professionals During the COVID-19 Pandemic in Poland
Brief Title: Clinical Trial Evaluating the Effect of BCG Vaccination on the Incidence and Severity of SARS-CoV-2 Infections Among Healthcare Professionals During the COVID-19 Pandemic in Poland
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hanna Czajka (Other)
Collaborators: Medical Research Agency, Poland (Other Government)
Responsible Party: Sponsor-Investigator, Hanna Czajka, National Project Coordinator, University of Rzeszow
Organization: University of Rzeszow (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: BCG/COVID-19/UR/04/2020; 2020-002111-22 (EudraCT Number)
Record Dates: First submitted 2020-10-18; First posted 2020-12-02 (Actual); Last update posted 2020-12-02 (Actual); Status verified 2020-11

CONDITIONS: Covid19; BCG Vaccination Reaction; SARS-CoV Infection
Keywords: Covid19; BCG Vaccination; SARS-CoV Infection; BCG vaccine
MeSH Terms: conditions — COVID-19; Severe Acute Respiratory Syndrome | interventions — Saline Solution

STUDY DESIGN:
Intervention Model Description: * Running the RT 23 test (visit No.2 - V2)
  * RT23 test reading and BCG -10 vaccination (visit No. 3-V3):
  Positive subjects:
  1. assigned to Group I, not randomised and not vaccinated against tuberculosis
  2. when the RT23 test indicates a strongly positive result /induration diameter > 15 mm/, the subject is informed to contact his/her family doctor to obtain a referral to a pulmonary outpatient clinic
  Negative subjects:
  1. undergo a physical examination before vaccination performed by the doctor (investigator)
  2. are remotely randomised by the e-CRF IT system to Group II receiving BCG-10 or to placebo Group III (control). The subject must not be informed about the group he/she belongs to receive BCG-10 or a placebo
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Due to trial blindness, the team (a doctor and nurse) participating in visits 2 (V2) and 3 (V3) (as unblinded staff) is excluded from further contacts with trial subjects and from participating in the trial.
  After the visit, the investigator enters its results into the medical documentation and the e-CRF system.
  In the medical records of visit 3 (written and electronic), the result of randomization is not disclosed.
  After visit 3, the division of subjects into Groups II and III (randomisation) is recorded only in separate written records; the physician participating in visit 2 and 3 sends the documentation to the leading centre after the end of visit 3, where it is stored and fully protected against access of blinded personnel.
  The subject must not be informed about the group he/she belongs to.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Group I (No Intervention): with positive RT23 test reading, not randomised and not vaccinated against tuberculosis
- Group II (Active Comparator): with negative RT23 test reading, receiving BCG-10 Vaccine
  Interventions: Drug: BCG-10 vaccine
- Group III (Placebo Comparator): with negative RT23 test reading, receiving placebo
  Interventions: Drug: 0.9% saline

INTERVENTIONS:
Drug: BCG-10 vaccine — The BCG-10 anti-tuberculosis vaccine
  * powder and solvent for preparing a suspension for intradermal injections of Vaccinum tuberculosis (BCG) cryodesiccatum;
  * lyophilised BCG vaccine
  * one dose (0.1 ml) contains 50 micrograms of half-dried mass of BCG mycobacteria, which corresponds to 150,000 - 600,000 of live BCG bacilli- the Brazilian Moreau sub-strain.
  Arms: Group II
Drug: 0.9% saline — 0.9% saline
  Arms: Group III

SUMMARY:
Countries that have not carried out universal mass vaccination against tuberculosis (BCG) have been shown to have higher incidence and death rates due to COVID-19 than countries with mass, long-term BCG immunization programmes.

The aim of the study is to answer the following questions:

1. Does BCG vaccination affect the course of COVID-19 (number of cases/deaths/severity of symptoms)?
2. Will the course of COVID-19 be milder among subjects with a negative TB skin test (PPD RT 23 SSI) after an additional dose of BCG than in case of non-vaccinated subjects?
3. Do people with a positive TB skin test have a milder course of COVID-19 infection than people with a negative test result?

A multicenter, randomized, partially blinded, placebo-controlled study will be conducted in Rzeszow/Krakow/ Katowice/Warsaw on a group of 1000 volunteers, health care workers according to the following schedule: V 0-1: inclusion/informed consent/interview; V2: administration of TB skin test/anti-SARS-CoV-2 IgG test/serum banking*; V3: TB skin test (TST) interpretation and subjects' division into three groups: (I) positive TST - observation; (II) negative TST- BCG-10 vaccination; (III) negative TST - placebo. Division into groups II and III based on randomisation; V4: serum banking*. Parallel beginning from V3, weekly telephone monitoring participants' health status; In case of COVID-19 symptoms a nasopharyngeal swab to confirm SARS-CoV-2 infection + serum banking*. V5: 3 months after vaccination at the end of the study: history/anti-SARS-CoV-2 IgG test, serum banking*.

Statistical analysis - comparison of the course of COVID-19 in groups: (I) with positive TST + observation, (II) with negative TST + BCG, (III) with negative TST + placebo - should demonstrate whether mass BCG vaccination has an impact on the incidence and course of COVID-19.

* to measure the level of cytokines involved in cell-mediated immunity process

DETAILED DESCRIPTION:
Trial design:

The multicentre, randomised, double-blind placebo-controlled trial will be conducted in five centres: Rzeszów, Kraków, Katowice, Warsaw (2 centres) in a group of 1000 volunteers, health care workers (physicians, nurses, midwives, paramedics, laboratory diagnosticians, electroradiology technicians, physiotherapists, nutritionists, and orderlies), both women and men aged ≥25 years and employed in health care facilities in the above-mentioned cities and provinces.

Planned duration of the trial:

2-4 weeks -recruitment, inclusion in the trial, RT 23 testing, BCG-10 vaccination 3 months - observation after vaccination 18 months, calculated from the date of trial initiation (visit no. "0"); during this period the subjects are to provide the Research Team with telephone information about possible hospitalisations and other unexpected, sudden or significant changes in health.

Recruitment period:

Sending invitations to participate in the trial to the healthcare professionals involved as well as providing the subjects with " Information for trial participants" leaflets and electronic "Informed Consent" forms

Inclusion in the trial (visit No.0 - V0):):

• obtaining informed consent to participate in the trial by exchanging electronic information and declarations of intent between the centre (investigator) and the individual declaring readiness to participate in research with double verification of the subject identity /e-mail+SMS/, which is intended to limit direct contacts during the period of COVID-19 epidemic risk

Inclusion in the trial (visit No.1 - V1):

* Investigator-subject telephone contact (in the days following V0 or directly during the same day)
* remote verification of the subject according to the inclusion and exclusion criteria, history taking regarding demographic characteristics, health status, and previous BCG vaccinations)
* setting the date of the RT23 test (place, day, time) to minimise the number of direct contacts between the research team and the subjects, in accordance with the current epidemic recommendations
* after the visit, the investigator enters the information obtained into the e-CRF system. The details concerning the visit and the scope of information collected are to be contained in V1 and V0/1 cards.
* after the visit, the investigator enters its results into the medical documentation and e-CRF system.

Running the RT 23 test (visit No.2 - V2):

* direct contact following the telephone contact to confirm the subject's health condition
* temperature measurement (non-contact thermometer), blood sampling (5 ml) for determinations of IgG SARS-CoV-2 antibodies and cytokine levels
* photographing the scars after BCG vaccination on the left forearm of the subject (without the details of appearance); the photographs are stored in the electronic documentation with the number assigned to a particular subject
* RT 23 trial initiation
* providing the subject with the written informed consent form, participant card, as well as the card of contacts, thermometer, and pregnancy test (females) in a sealed plastic envelope
* the visit will be carried out in accordance with the procedures in force in departments of infectious diseases
* setting the date (date and time) of the third visit- after 72 hours
* after the visit, the investigator will enter its results into the medical documentation and e-CRF system.

RT23 test reading and BCG -10 vaccination (visit No.3-V3)

* the direct visit, preceded by the telephone contact to confirm the subject's health status
* before the visit, the female subjects perform a pregnancy test in the morning hours; those with positive results are excluded from the trial
* temperature measurement (non-contact thermometer)
* the visit will be carried out in accordance with the procedures in force in departments of infectious diseases.
* reading of the tuberculin test run during visit 2 (according to the criteria) and photographing the post-test induration on the left arm of the subject (for documentation purposes), no appearance details; the photos are stored in the electronic documentation marked with the number given to a particular study subject.

Positive subjects:

* are assigned to Group I, are not randomised and are not vaccinated against tuberculosis
* are subjected to a weekly remote medical follow-ups in agreement with the "telephone contact card" until the trial completion (3 months from the date of visit 3 of the last subject); the follow ups are conducted by the investigator, a member of the research team, not participating in visit 3;
* when the RT23 test indicates a strongly positive result /induration diameter > 15 mm/, the subject is informed to contact his/her family doctor to obtain a referral to a pulmonary outpatient clinic.

Negative subjects:

* undergo a physical examination before vaccination performed by the doctor (investigator)
* are remotely randomised by the e-CRF IT system to Group II receiving BCG-10 or to placebo Group III (control). The subject must not be informed about the group he/she belongs to
* receive BCG-10 or a placebo in intradermal injections performed by a trained nurse with appropriate professional experience
* undergo weekly remote medical observations carried out by the investigator not involved in visit 3, according to the "telephone contact card", until the trial completion (3 months from the date of visit 3 of the last subject) Due to trial blindness, the team (a doctor and nurse) participating in visits 2 (V2) and 3 (V3) (as unblinded staff) is excluded from further contacts with trial subjects and from participating in the trial.

After the visit, the investigator enters its results into the medical documentation and the e-CRF system.

In the medical records of visit 3 (written and electronic), the result of randomization is not disclosed.

After visit 3, the division of subjects into Groups II and III (randomisation) is recorded only in separate written records; the physician participating in visit 2 and 3 sends the documentation to the leading centre after the end of visit 3, where it is stored and fully protected against access of blinded personnel.

Blood collection - visit No. 4 (V4):

* within 6-8 weeks after visit 3, all subjects are invited by telephone to the place designated by the Principal Investigator to take 5 ml blood samples to determine the levels of cytokines
* blood collection is carried out by a member of the research team appointed by the Principal Investigator
* after the visit, the investigator enters its results into the e-CRF system.

Blood collection - visit No. 5 (V5):

* three months after visit 3, all subjects are invited by telephone to the place designated by the Principal Investigator to take 5 ml blood samples to determine SARS-CoV-2 IgG antibodies and cytokine levels
* blood collection is carried out by a member of the research team appointed by the Principal Investigator
* after the visit, the investigator enters its results into the medical documentation and the e-CRF system.

Remote phone visit

• carried out for a period of three months between visit 3 (V3) and visit 5 (V5), once a week; during this visit the physician (member of the research team) asks questions according to the attached phone contact card.

Interventional visit

* will be carried out between visit 3 and visit 5, when the symptoms determined in the telephone Contact card appear to indicate a possible SARS-CovV-2 infection.
* the trial subject contacts by telephone the investigator conducting a weekly remote medical observation, and if the score 3 is obtained during the telephone evaluation of health, the mobile team is deployed to the subject
* the ambulance takes a swab from the subject's nasopharynx and collects 5 ml of blood for cytokine determinations to confirm the infection with this virus or otherwise. The visit will be carried out at the subject's place of residence and the material collected will be delivered to a respective analytical laboratory
* after the visit, the investigator will enter its results into the medical documentation and the e-CRF system

Moreover,

* each subject may contact the research centre by phone 24 hours a day, 7 days a week
* each subject may withdraw from the trial at any time.
* when the telephone contact with the subject is infeasible, the research team may use the reserve contact indicated by the subject or contact the hospital attending the subject
* if the subject develops the symptoms of COVID-19 during the trial, he/she has to adhere to the generally applicable rules
* at the end of the study, all subjects in groups II and III will be notified (individually and confidentially) whether they have received BCG-10 or placebo
* when a preliminary result indicates the significant benefits of additional BCG vaccination, an additional dose of BCG-10 will be offered to all non-vaccinated subjects.

Statistical analysis Statistical analysis will be conducted using MedCalc v17.7 software. The quantitative variables will be presented as an arithmetic mean and standard deviation (variables with a normal distribution) or median and interquartile range (variables with a non-normal distribution/ a skewed distribution). The distribution will be assessed using the Shapiro-Wilk test. The qualitative variables will be presented as an absolute value and percentage. The inter-group differences for quantitative variables will be evaluated by the Student's t-test or analysis of variance (independent samples, variables with a normal distribution), and the Mann-Whitney U or Kruskal-Wallis test (independent samples, skewed variables).

In cases where significant inter-group differences have been demonstrated based on the ANOVA or Kruskal-Wallis test, a post-hoc analysis will be performed. The significance of differences for quantitative dependent variables will be assessed applying the Student t-test for dependent samples or the non-parametric equivalent of variance analysis, or the Wilcoxon signed-rank or Friedman's rank test (depending on the number of groups and the distribution). For unrelated qualitative variables, the chi-squared test or Fisher's exact test will be used, while for related variables the McNemar's test will be applied. The correlation between inter-qualitative variables will be analysed using the Pearson correlation analysis or Spearman's rank correlation. For selected qualitative dependencies for quality dichotomous variables, the odds ratios (or relative risk factors) and their 95% confidence intervals will be calculated. The results of simple analyses will be the basis for advanced statistical analysis methods, i.e. logistic regression models or multiple regression analyses. Models will include variables with p<0.1 in simple analysis will be included in the models mentioned above. Moreover, the odds ratios together with 95% confidence intervals (logistic regression) or regression coefficients with their standard error (multiple regression) will be estimated. Finally, p<0.05 will be considered statistically significant.

Minimum number of trial subjects:

A/ Assuming that 50% of individuals have negative tuberculin test results when alpha=0.05 and measurement precision=5%, a group of at least 384 subjects (~400) should be recruited. Assuming a 10 % loss of subjects between the initiation and reading of the tuberculin test, the group subjected to the tuberculin test should contain at least 450 people.

B/ Assuming a 10% difference in endpoint occurrence (disease) when alpha=0.05 is expected, at least 193 individuals in each group (~200) should be examined. Given the loss to follow -up of 10 %, each group (study and control) should include at least 220 individuals.

C/ In conclusion, considering all the above calculations, at least 880 individuals (~900) should be included in the trial. Given that 10% of subjects will not give their informed consent to participate in the trial, at least 990 individuals (~1000) should be invited to the project.

Note: Six weeks after the inclusion of the last subject, the number of serious adverse events (SAEs) in each group is to be analysed in order to decide whether to continue the follow-up or to administer the BCG vaccine to all non-vaccinated subjects.

Data analysed:

1. Incidence and deaths rates in the study group
2. Additionally:

   * documented SARS-CoV-2 infection
   * duration of symptoms
   * types of symptoms and their frequency
   * average duration of domestic isolation
   * maintenance of body temperature ≥37.5oC, in the ranges of:

     1. 37.5C-38.0C
     2. 38.1C-39.0C
     3. more than 39C
   * in the case of hospitalisation: length of treatment, including possible ICU stay, ventilator therapy, complications, death.
3. group characteristics:

   * date of inclusion (date of signing informed consent to participate in the trial)
   * age (month, year of birth)
   * gender
   * body weight, height, BMI
   * province of residence (Podkarpackie, Małopolska, Silesian, Mazovian)
   * workplace (department, ER, outpatient clinic, analytical laboratory)
   * profession (physician, nurse, midwife, paramedic, laboratory diagnostician, nutritionist, electroradiology technician, physiotherapist, orderly)
   * working hours per month, number of jobs during the pandemic
   * shift work (YES/NO)
   * percentage of hours of direct contact with the patient (four intervals <25%, 25-50%, 50-75%, >75%)
   * cardiovascular diseases: hypertension, ischaemic heart disease, post-myocardial infarct condition, atrial fibrillation, chronic heart failure, others - which ones?
   * respiratory diseases: asthma, chronic obstructive pulmonary disease (COPD), interstitial lung disease, others- which ones?
   * diseases of the nervous system: epilepsy, post-stroke condition, polyneuropathy, others- which ones?
   * diseases of the osteoarticular system: osteoarthritis, rheumatoid arthritis, others- which ones?
   * diseases of the gastrointestinal system: liver diseases - list them, bowel diseases- list them, pancreatic diseases- list them, others: which ones?
   * kidney disease: chronic kidney disease, kidney stones, others- which ones?
   * diabetes: type 1; type 2: diet/insulin?
   * autoimmune diseases: which ones?
   * other chronic diseases: which ones?
   * neoplastic diseases: which ones? how treated? when?
   * smoking: pack-year? E-cigarettes: years?
   * allergies: which ones?
   * BCG vaccinations to this day.

Laboratory tests during the trial:

1. standard planned blood test during visit 2 (running the RT23 test,) -collection of 5 ml of blood (determination of the presence of SARS-CoV-2 IgG antibodies, determination of the level of cytokines regulating cellular immunity - hereinafter referred to as the cytokine level)
2. within 6-8 weeks after BCG vaccination, collection of 5 ml of blood for cytokine level determinations
3. after the completion of follow-ups (3 months after the last study participant was included), collection of 5 ml of blood (for determination of IgG antibody levels, SARS-CoV-2 virus, and cytokine levels).
4. if COVID-19 symptoms occur in the subject:

   1. the subject eligible for hospitalisation will be urgently (emergently) hospitalised due to COVID-19 and tested according to the procedures in force in the hospital; moreover, each subject will receive an identifier (similar to ID) with information about participation in the trial and a request to the personnel assuming care of the subject to inform the research team and secure samples (5 ml of blood for cytokine determination and a swab from the nasopharynx for the SARS-CovV-2 genetic material testing)
   2. in the case of the subject not eligible for hospitalisations with symptoms suggestive of the infection but not requiring hospitalisation, symptoms and their duration will be noted and during the intervention visit 5 ml of blood will be sampled for cytokine determinations and a nasopharyngeal swab will be taken for testing whether SARS-CoV-2 genetic material is present or otherwise. The material will be collected at the subject's home in accordance with the safety procedure.

      Methodology of laboratory tests Laboratory blood tests for determinations of SARS-CoV-2 IgG antibodies and cytokine levels will be carried out..

      Procedure - collection and transport of material to the laboratory preparing it for banking

      • Collection of nasopharyngeal swabs for SARS CoV-2 genetic material testing using the RT-qPCR test and blood sampling to assess cytokine and/or IgG levels

      Criteria for completion of the trial

      According to its program, the trial will last for a period of 3 months from the date of visit No. 3 (administration of the vaccine) to the date of visit 5 (blood collection for determinations of IgG SARS-CoV-2 antibodies and cytokine levels).

      Over the next 15 months, the subjects will be asked to provide the Research Team with telephone information about possible hospitalizations and other unexpected, sudden or significant changes in their health.

      The trial will be completed after the last visit of the last subject and after the results serological and genetic tests (PCR-SARS) are available, approximately 8 months after its initiation.

      The observation of possible SAEs reported by the subjects will be completed 18 months after the commencement of the trial.

ELIGIBILITY:
Inclusion Criteria:

* a health care professional (physician, nurse, midwife, paramedic, electroradiology technician, laboratory diagnostician, physiotherapist, nutritionist, orderly) aged >25 years
* no confirmed SARS-CoV-2 infection
* informed consent to participate in the trial and consent to personal data processing
* declared availability for telephone contacts throughout the study period
* good health condition
* earlier vaccination against tuberculosis

Exclusion Criteria:

* hypersensitivity to any component of BCG-10
* hypersensitivity to previously administered tuberculin (local skin lesions, necrosis of the skin, blisters, other severe skin reactions at the injection site)
* HIV infection (confirmed or suspected infections, even if they are asymptomatic)
* primary or secondary immunodeficiencies (including interferon - gamma deficiency or DiGeorge syndrome)
* radiotherapy (less than 24 months before the date of inclusion in the trial
* treatment with corticosteroids, ongoing immunosuppressive therapy (including those treated with monoclonal antibodies to TNF-α, such as infliximab) - less than 24 months before the date of inclusion in the trial
* neoplastic diseases (e.g. leukaemia, malignant granuloma, lymphoma or some other cancer of the reticuloendothelial system) - less than 24 months before the date of inclusion in the study
* after stem cell transplantation and organ transplantation
* in the exacerbation stage of chronic diseases (including severe malnutrition)
* pregnancy
* history of tuberculosis
* keloid at the vaccination site after previous BCG vaccination

Min Age: 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2020-07-07 (Actual); Primary Completion 2020-12 (Estimated); Study Completion 2021-04 (Estimated)

PRIMARY OUTCOMES:
death and life- or health-threatening condition (cardiac arrest with effective resuscitation, shock, severe respiratory failure, severe renal failure, stroke/transient cerebral ischaemia) | throughout the period of 18 months from inclusion
  * shock - when catecholamines are required despite initial fluid resuscitation
  * severe respiratory failure - the need for non-invasive or invasive ventilation
  * severe renal failure - the need for renal replacement therapy (for undialysed individuals, i.e. with end-stage renal failure (ESRD)

SECONDARY OUTCOMES:
Onset of clinical symptoms of COVID-19 | 12 weeks from the date of the third visit - V3
  Present symptoms (determined in the Telephone Contact Card) appear to indicate a possible SARS-CovV-2 infection
asymptomatic SARS-CovV-2 infection | 12 weeks from the date of the third visit - V3
  based on anti SARS-CoV-2 IgG serological tests
Hospitalisation | 12 weeks from the date of the third visit - V3
  the need for hospitalisation and its duration
ICU Hospitalisation | 12 weeks from the date of the third visit - V3
  the need for hospitalisation in the ICU and its duration
Dyspnoea | 12 weeks from the date of the third visit - V3
  requiring passive oxygen therapy to eliminate the symptom or maintain saturation >92%

CONTACTS AND LOCATIONS:
Overall Officials: Hanna Czajka, prof., Principal Investigator — College of Medical Sciences, University of Rzeszów
Locations (6):
- Poland (6):
  - Department of Anesthesiology and Intensive Care, University Clinical Center, School of Medicine in Katowice, Medical University of Silesia, Katowice
  - Stefan Żeromski Specialist Hospital, Krakow
  - Voivodeship Hospital nr 2 in the Name of The Saint Queen Jadwiga, University of Rzeszów, Poland, Rzeszów
  - Saint Jadwiga Śląska Hospital, Trzebnica
  - Department of Pediatrics, Bielanski Hospital,, Warsaw
  - Praski Hospital, Warsaw

IPD SHARING:
Plan to Share IPD: Undecided